CLINICAL TRIAL: NCT04431141
Title: A Randomized, Open-label, Multiple-dose, Cross-over Dosing Study to Evaluate Pharmacokinetic Drug Interaction Between Teneligliptin and Empagliflozin in Healthy Adults
Brief Title: Pharmacokinetic Drug Interaction Between Teneligliptin and Empagliflozin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Handok Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MP-C105
Record Dates: First submitted 2020-06-04; First posted 2020-06-16 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 3-(4-(4-(3-methyl-1-phenyl-1H-pyrazol-5-yl)piperazin-1-yl)pyrrolidin-2-ylcarbonyl)thiazolidine; empagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Teneligliptin (Experimental)
  Interventions: Drug: Teneligliptin
- Empagliflozin (Experimental)
  Interventions: Drug: Empagliflozin
- Teneligliptin and Empagliflozin (Experimental)
  Interventions: Drug: Teneligliptin and Empagliflozin

INTERVENTIONS:
Drug: Teneligliptin — Teneligliptin alone
  Other Names: Tenelia®
  Arms: Teneligliptin
Drug: Empagliflozin — Empagliflozin alone
  Other Names: Jardiance®
  Arms: Empagliflozin
Drug: Teneligliptin and Empagliflozin — Teneligliptin and empagliflozin
  Other Names: Tenelia® and Jardiance®
  Arms: Teneligliptin and Empagliflozin

SUMMARY:
This study is to evaluate pharmacokinetic drug interaction between teneligliptin and empagliflozin in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults between 19 and 45 years of age (both inclusive) at the screening visit
* Body mass index between 19 kg/m2 and 28 kg/m2 (both inclusive) at the screening visit
* Subjects must voluntarily decide to participate in the study and provide written informed consent to comply with study instructions

Exclusion Criteria:

* History of type 1 diabetes mellitus and/or diabetic ketoacidosis
* Severe infection, surgery, or severe trauma within 6 months prior to the screening visit
* Hereditary problems such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
* Treatment with any investigational product or study drug in another clinical trial or bioequivalence study within 180 days prior to the screening visit
* Any laboratory test or 12-lead ECG finding based on which the subject is determined ineligible to participate in the study
* Subject determined by the principal investigator to be ineligible for study conduct for other reasons

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2020-11-16 (Actual); Study Completion 2021-01-25 (Actual)

PRIMARY OUTCOMES:
Cmax,ss of teneligliptin and empagliflozin | 72 hours
  Peak Plasma Concentration (Cmax) at steady state
AUCτ,ss of teneligliptin and empagliflozin | 72 hours
  Area under the plasma concentration versus time curve (AUC) at steady state

SECONDARY OUTCOMES:
Tmax,ss of teneligliptin and empagliflozin | 72 hours
  Time to reach Cmax,ss
t1/2β of teneligliptin and empagliflozin | 72 hours
  Terminal elimination half-life

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Pharmacology, Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No